CLINICAL TRIAL: NCT00199433
Title: A Phase 2, Double-blind, Placebo-controlled, Randomized, Parallel-Group, Multicenter Study to Evaluate the Efficacy and Safety of 40mg/Day KW-6002 (Istradefylline) as Monotherapy in Subjects With Parkinson's Disease
Brief Title: A Study of Istradefylline (KW-6002) as Monotherapy in Parkinson's Disease (PD) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin, Inc. (Industry)
Collaborators: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6002-US-051
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Parkinson's Disease; Movement Disorder Syndrome
Keywords: Parkinson's Disease; Movement Disorder; Neurology,; Clinical Trial
MeSH Terms: conditions — Parkinson Disease; Movement Disorders | interventions — istradefylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Istradefylline (KW-6002)

SUMMARY:
The primary purpose of this study is to evaluate the efficacy, safety, and tolerability of 40 mg per day of istradefylline (KW6002) as monotherapy in patients with Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's disease is a progressive disease which results in deterioration of motor function and is the result of dopamine depletion in specific brain structures. Current therapeutic approaches include dopamine replacement and the use of dopamine receptor agonist drugs. These therapies are effective but may be associated with unwanted complications like wearing off phenomena and involuntary abnormal movements (dyskinesia). Istradefylline may provide a nondopaminergic approach to the treatment of Parkinson's disease.

This study will compare the efficacy of 40 mg per day of istradefylline in improving the symptoms of Parkinson's disease with placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Early PD by UKPDS criteria
2. Mild to moderate difficulty daily activities
3. Females: Either postmenopausal or willing to use adequate contraception

Exclusion Criteria:

1. Unable to discontinue current PD medication
2. Exposure to Levodopa for more than 1 month
3. Symptoms that may suggest a diagnosis other than Parkinson's disease
4. Medical conditions and/or abnormal laboratory findings which preclude participation including cancer in the last 5 years, a history of drug abuse/dependence, abnormal cognitive status, a history of seizures, neuroleptic malignant syndrome, psychosis, or abnormal liver function tests

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2005-05; Primary Completion 2006-07 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the UPDRS subscale III at endpoint.

SECONDARY OUTCOMES:
Interim actual and change from baseline values in UPDRS total and subscale scores, Clinical Global Impression, measures of motor performance, and neuropsychological testing.
Safety:
Exam
vitals
weight
ECG
laboratory tests and adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Neil Sussman, MD, Study Director — Kyowa Kirin, Inc.
Locations (1):
- Kyowa Pharmaceutical Inc., Princeton, New Jersey, United States